CLINICAL TRIAL: NCT07122661
Title: STudy of Real World vaccinE Effectiveness of maTernal RSVpreF vaccinatiON Against Respiratory Syncytial Virus (RSV) in Hospitalised Infants in Australia
Brief Title: STudy of Real World vaccinE Effectiveness of maTernal RSVpreF vaccinatiON Against Respiratory Syncytial Virus (RSV) in Hospitalised Infants in Australia (STREETON)
Acronym: STREETON
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: The Kids Research Institute Australia on behalf of the Centre for Child Health Research, University of Western Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: C3671066
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus (RSV); Respiratory Syncytial Virus; Lower Respiratory Tract Disease; Respiratory Tract Diseases; Acute Respiratory Illness (ARI)
Keywords: RSVpreF; Vaccine; Effectiveness; Vaccine Effectiveness; Pregnancy; Maternal; Immunization; Maternal Immunization; ABRYSVO; Respiratory Syncytial Virus; Lower Respiratory Tract Disease; Infants; Hospitalized; Hospitalization; Test Negative Design; Case Control; Retrospective; Respiratory Outcomes; Prefusion F protein-based; Acute Respiratory Illness
MeSH Terms: conditions — Respiratory Tract Diseases | interventions — abrysvo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Infants who meet the respiratory clinical case definition and test positive for RSV (result obtained from standard of care testing with specimen collected within 10 days prior to hospital admission through 3 days after a hospital admission).
  Interventions: Biological: ABRYSVO
- Controls: Infants who meet the respiratory clinical case definition and test negative for RSV (result obtained from standard of care testing with specimen collected within 10 days prior to hospital admission through 3 days after a hospital admission).
  Interventions: Biological: ABRYSVO

INTERVENTIONS:
Biological: ABRYSVO — This is a non-interventional retrospective study; therefore, ABRYSVO vaccine has already been administered according to the standard of care. ABRYSVO is a bivalent RSV prefusion F protein-based vaccine (RSVpreF) composed of two prefusion F proteins to protect against both RSV-A and RSV-B.
  Other Names: RSVpreF; RSV Prefusion F

SUMMARY:
This Pfizer-sponsored real-world retrospective non-interventional study will be conducted within a research network comprised of independent hospitals across Australia using data collected during routine standard of care clinical encounters available in health records, supplemented with information from the official national immunisation registry, the Australian Immunisation Register. Additional data from accredited pathology laboratories will be included. There will be no active enrollment of study participants, no direct contact with study participants, and no collection of any primary data outside of the standard of care.

This study will use a test negative design to evaluate real-world vaccine effectiveness of RSVpreF vaccination during pregnancy against RSV-associated outcomes in infants.

DETAILED DESCRIPTION:
This case-control study using a test negative design will include all infants through 12 months of age who were admitted to one of the participating hospitals with symptoms of respiratory infection, met the clinical case definition of acute respiratory illness, and had a respiratory specimen collected within 10 days prior to hospital admission through 3 days after a hospital admission with an RSV test result through standard of care testing.

The primary objective is to estimate vaccine effectiveness (VE) of ABRYSVO during pregnancy against RSV-positive lower respiratory tract disease (LRTD) hospitalisation among infants from birth through 6 months (0 to ≤180 days) of age.

Baseline characteristics of the study population will be described by case/control status and by maternal RSVpreF vaccination status. Standardised mean differences may be used to compare the distributions (absolute differences >0.10 will be considered meaningful). For all VE objectives, we will use a logistic regression model to compare the odds of maternal ABRYSVO vaccination during pregnancy between test-positive cases and test-negative controls, generating an odds ratio (OR) and 95% CI and we will use multivariable logistic regression to compute an adjusted OR (aOR), from which we will derive final VE estimates, adjusted for potential confounding, according to the formula: VE = (1-aOR) x 100%.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Infant ≤12 months (≤360 days) of age on the hospitalisation date.
2. Index date within the time period for data collection (approximately 01 March 2025 - 28 February 2027)
3. Hospitalised with acute respiratory illness meeting the protocol-defined clinical case definition, and for whom RSV testing results from a specimen collected 10 days prior to hospital admission through 3 days after a hospital admission are known.
4. Infant born to a birth mother eligible to receive ABRYSVO vaccination, with infant date of birth on or after 17 February 2025.

Exclusion Criteria:

Participants meeting any of the following criteria will not be included in the study:

1. Infant born at <28 weeks and 0/7 days of gestational age.
2. Infant received any licensed or investigational RSV preventive product (e.g., palivizumab, nirsevimab, active RSV vaccine) since birth.
3. Infant received ≥1 blood transfusion or other blood products containing antibody (e.g., fresh frozen plasma) since birth.
4. Infant born to a birth mother who received any other licensed or investigational RSV vaccine during this pregnancy.
5. Infant born to a birth mother for whom ABRYSVO vaccination status cannot be confirmed in available data sources.

Ages: 0 Years to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This hospital-based retrospective study will be conducted in up to 9 hospitals across 6 states/territories in Australia, supported by the Paediatric Active Enhanced Diseases Surveillance Network.
  Given the retrospective nature of this study, hospitals that already function as national sentinel units for respiratory virus surveillance, or have robust clinical, laboratory or epidemiological surveillance will be included. Each participating hospital conducts year-round standard of care testing for acute respiratory illness which includes respiratory virus panel test using PCR.
  Study will include all infants through 12 months of age who were admitted to one of the participating hospitals with symptoms of respiratory infection, met the clinical case definition of acute respiratory illness, and had a respiratory specimen collected within 10 days prior to hospital admission through 3 days after a hospital admission with an RSV test result through standard of care testing.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Estimate vaccine effectiveness of ABRYSVO during pregnancy against RSV-positive lower respiratory tract disease hospitalisation among infants. | From birth through 6 months (0 to ≤180 days) of age.
  RSV-positive lower respiratory tract disease hospitalisation occurring 0 to ≤180 days after birth.

SECONDARY OUTCOMES:
Estimate vaccine effectiveness of ABRYSVO during pregnancy against RSV-positive lower respiratory tract disease hospitalisation among infants. | From birth through 6 months (0 to ≤180 days) of age within key subgroups.
  RSV-positive lower respiratory tract disease hospitalisation occurring 0 to ≤180 days after birth subgrouped by:
  * gestational age at ABRYSVO vaccination.
  * gestational age at birth.
  * time from ABRYSVO vaccination to birth.
  * time intervals of infant age at illness, including cumulative (e.g., 0 to ≤3 months, 0 to ≤6 months) and discrete (e.g., 0 to ≤3 months, >3 to ≤6 months) age intervals.
Estimate vaccine effectiveness of ABRYSVO during pregnancy against RSV-positive severe lower respiratory tract disease hospitalisation among infants. | From birth through 6 months (0 to ≤180 days) of age and within key subgroups.
  RSV-positive lower respiratory tract disease hospitalisation occurring 0 to ≤180 days after birth subgrouped by:
  * gestational age at ABRYSVO vaccination.
  * gestational age at birth.
  * time from ABRYSVO vaccination to birth.
  * time intervals of infant age at illness, including cumulative (e.g., 0 to ≤3 months, 0 to ≤6 months) and discrete (e.g., 0 to ≤3 months, >3 to ≤6 months) age intervals.
Estimate vaccine effectiveness of ABRYSVO during pregnancy against RSV-positive acute respiratory illness hospitalisation among infants. | From birth through 6 months (0 to ≤180 days) of age and within key subgroups.
  RSV-positive acute respiratory illness hospitalisation occurring 0 to ≤180 days after birth subgrouped by:
  * gestational age at ABRYSVO vaccination.
  * gestational age at birth.
  * time from ABRYSVO vaccination to birth.
  * time intervals of infant age at illness, including cumulative (e.g., 0 to ≤3 months, 0 to ≤6 months) and discrete (e.g., 0 to ≤3 months, >3 to ≤6 months) age intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.